CLINICAL TRIAL: NCT00714649
Title: Neoadjuvant Cetuximab Monotherapy Followed by Surgery in Squamous Cell Carcinoma of Head and Neck: Phase I/II Study
Brief Title: Neoadjuvant Cetuximab in HNSCC Combined With Curative Surgery
Acronym: CHIRON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Merck Serono International SA (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIRON 2008-01
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Carcinoma treated with surgery; and/or radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-1 (Other): This is a phase I/II trial. PhaseI: The delay between the last administration of cetuximab and surgery will be progressively reduced. Five delay schedules are pre-defined before final administration of 3 preoperative doses of cetuximab with a 24-hour delay between the last dose of cetuximab and surgery. The cohort size is 3 patients per delay schedule, extended to 6 patients if one "limiting toxicity" is observed.
  Phase II: will proceed if delay schedule V is safe. The patients included in delay schedule V of the Phase I part of the study will be involved in the phase II analysis. Recruitment of a total of 12 patients (3-6 of delay schedule V in phase I plus an additional 3-9 patients).
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — Cetuximab 250mg/m²/week IV before surgery till surgery

SUMMARY:
Primary diagnose HNSCC carcinoma patients eligible for curative surgery will be proposed the addition of 2 or 3 neoadjuvant cetuximab infusions. The main objective is to reduce to a minimal delay the time elapsing between last infusion and surgery.

Iterative biomarkers will be taken at 6 time points permitting to investigate expression gen profile and protein mutation.

DETAILED DESCRIPTION:
This is a Phase I/II trial of neoadjuvant cetuximab monotherapy in the preoperative treatment of patients with operable HNSCC. It is a monocenter study (St-Luc university Hospital, Université catholique de Louvain, Brussels).

This part of the trial will determine the safe minimum delay between the neoadjuvant cetuximab infusion and surgery. The aim is to investigate if cetuximab given 24 hours before surgery is safe.

Patients will receive cetuximab with a loading dose of 400 mg/m2 for the first administration followed by 250 mg/m2/week at the second and third administrations, if applicable. The delay between the last administration of cetuximab and surgery will be progressively reduced (Figure 1).

Five levels are pre-defined before final administration of 3 preoperative doses of cetuximab with a 24-hour delay between the last dose of cetuximab and surgery.

Level I: 10-12 days delay between the second cetuximab infusion and surgery (total of 2 doses pre-op) Level II: 6-8 days delay between the second cetuximab infusion and surgery (total of 2 doses pre-op) Level III: 3-4 days delay between the second cetuximab infusion and surgery (total of 2 doses pre-op) Level IV: 3-4 days delay between the third cetuximab infusion and surgery (total of 3 doses pre-op) Level V: 24-hour delay between the third cetuximab dose and surgery (total of 3 doses pre-op) The cohort size is 3 patients per level, extended to 6 patients if one "limiting toxicity" is observed. Decision rules are the same than as in any classic 3+3 phase 1design (Figure 2).

"Limiting toxicity" is defined as (i) any life-threatening (grade 4) surgical complication or (ii) an unexpected surgical grade 3 toxicity. Unexpected toxicity will be determined by the safety committee after careful review of the patient file.

The safety committee will consist of the surgical team of UCL Saint-Luc, one external surgeon, one representative from Merck and the study coordinators.

Patients treated at level V will be evaluated like patients in the phase II part.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* Histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx
* patients selected for a primary surgical treatment
* No distant metastases
* No active second malignancy during the last 5 years
* No prior or concurrent evidence of uncontrolled severe pathology precluding administration of surgery
* life expectancy more than 3 months
* Not pregnant or nursing; fertile patients both male or female, must use effective contraception
* Signed informed consent
* Performance Status ECOG 0-1

Exclusion Criteria:

* Nasopharynx cancer
* Past or current malignancy other than HNSCC
* performance Status ECOG above 2
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Use of any investigationals agents within 4 weeks prior ti entry
* Previous exposure to EGFR targeting therapy
* Known grade hypersensitivity to cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To investigate the safety administration of cetuximab - Phase 1: to determine the safe minimum delay between preoperative cetuximab infusion and surgery -Phase II: to investigate the safety of the minimum delay determined in the phase I part. | 10 weeks

SECONDARY OUTCOMES:
To investigate the safety of postoperative radiation therapy in combination with cetuximab | 10 weeks
To investigate the efficacy of cetuximab monotherapy in the pre-operative setting, using FDG-PET and PET/CT scan. | 10 weeks
To perform translational research | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal H Machiels, MD PhD, Principal Investigator — Cliniques Universitaires St Luc-UCL
Locations (1):
- Cliniques Universitaires St Luc-UCL, Brussels, Belgium